CLINICAL TRIAL: NCT03380676
Title: Study of Speech Disorders , Voice and Swallowing in Primary Dystonia Oromandibular
Acronym: DOM
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_34; 2013-A01299-36 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-11-08; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Dystonia, Primary; Dysarthria; Dysphonia; Dysphagia
MeSH Terms: conditions — Dystonic Disorders; Dysarthria; Dysphonia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oromandibular dystonia group: Patients with idiopathic oromandibular dystonia, either focal or associated to other dystonic features including generalized dystonia
- Healthy subjects: Healthy subjects (normal neurological examination), each being age-matched to a subjet of the oromandibular dystonia group

SUMMARY:
To better define the clinical characteristics of oromandibular dystonia, we aimed to study voice, speech and swallowing disorders in idiopathic oromandibular We planned to include consecutive patients followed in Lille Movement disorders department for idiopathic oromandibular dystonia and matched, healthy control subjects. Voice and speech disorders had to be assessed with the phonetic analysis, perceptive analysis and motor examination modules of the "Batterie d'Evaluation Clinique de la Dysarthrie" (Clinical Evaluation of Dysarthria), the Grade, Rough, Breathy, Asthenic, Strained scale, and a computer recording. Activities of daily living had to be assessed with the Oromandibular Dystonia Questionnaire, the Voice Handicap Index and the Deglutition Handicap Index.

ELIGIBILITY:
Inclusion Criteria:

* Both groups: Man or woman Age > 18 years French social security French speaking: fluent
* Oromandibular dystonia group: Idiopathic oromandibular dystonia (focal or associated to other dystonic symptoms)
* Healthy controls group: Same age +/- 2 years than a patient from the oromandibular dystonia group Normal clinical examination

Exclusion Criteria:

* Both groups: Any pathology making the orthophonic evaluation difficult Property protection regime Deprivation of liberty -Oromandibular dystonia group: Abnormal neurological examination, except dystonic features
* Healthy controls group: History of brain lesion Abnormal neurological examination Swallowing difficulties

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Oromandibular dystonia group
  * Healthy controls group
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
French scale "Batterie d'Evaluation Clinique de la Dysarthrie" (Clinical Evaluation of Dysarthria) phonetic analysis. | 10 minutes at baseline
  To describe the clinical characteristics of dysarthria in idiopathic oromandibular dystonia. Composite score (min=best=0; max=worst=151) including three subscales: phonetic production (min=worst=0; max=best=33); simple words (min=worst=0; max=best=88); complex words (min=wost=0; max=best=30).

SECONDARY OUTCOMES:
French software "Logiciel d'Evaluation Vocale Assistée" (Computer-Assisted Voice Assessment): maximum phonation time | 1 minute at baseline
  To describe the clinical characteristics of voice impairment in idiopathic oromandibular dystonia. Maximum phonation time was measured in seconds.
French software "Logiciel d'Evaluation Vocale Assistée" (Computer-Assisted Voice Assessment): frequency variations | 1 minute at baseline
  To describe the clinical characteristics of voice impairment in idiopathic oromandibular dystonia. Frequency variations were measured in Hz.
French software "Logiciel d'Evaluation Vocale Assistée" (Computer-Assisted Voice Assessment): number of pauses. | 1 minute at baseline
  To describe the clinical characteristics of voice impairment in idiopathic oromandibular dystonia. The number of pauses was counted.
French software "Logiciel d'Evaluation Vocale Assistée" (Computer-Assisted Voice Assessment): total lecture time. | 1 minute at baseline
  To describe the clinical characteristics of voice impairment in idiopathic oromandibular dystonia. Total lecture time was measured in seconds.
French software "Logiciel d'Evaluation Vocale Assistée" (Computer-Assisted Voice Assessment): pauses duration | 1 minute at baseline
  To describe the clinical characteristics of voice impairment in idiopathic oromandibular dystonia. Pauses duration was measured in seconds.
French software "Logiciel d'Evaluation Vocale Assistée" (Computer-Assisted Voice Assessment): fundamental frequency | 1 minute at baseline
  To describe the clinical characteristics of voice impairment in idiopathic oromandibular dystonia. Fundamental frequency was measured in Hz
French software "Logiciel d'Evaluation Vocale Assistée" (Computer-Assisted Voice Assessment): repetitions. | 2 minutes at baseline
  To describe the clinical characteristics of voice impairment in idiopathic oromandibular dystonia. Repetitions were measured in seconds.
French software "Logiciel d'Evaluation Vocale Assistée" (Computer-Assisted Voice Assessment): mean vocal intensity | 1 minute at baseline
  To describe the clinical characteristics of voice impairment in idiopathic oromandibular dystonia. Mean vocal intensity was measured in dB
Voice handicap index | 10 minutes at baseline
  To describe impairment of daily living activities in idiopathic oromandibular (min=best=0; max=worst=120)
Tohara swallowing test | 5 minutes at baseline
  To describe the clinical characteristics of swallowing difficulties in idiopathic oromandibular dystonia. Min=best=0; max=worst=4
Deglutition Handicap Index | 10 minutes at baseline
  To describe impairment of daily living activities in idiopathic oromandibular dystonia. Qualitative: 30 questions (possible answers: never; almost never; sometimes; often; always)
Oromandibular dystonia questionnaire | 10 minutes at baseline
  To describe impairment of daily living activities in idiopathic oromandibular dystonia. Qualitative: 25 questions (possible answers: never; almost never; sometimes; often; always)
Grade Rough Breathy Asthenic Strained scale | 5 minutes at baseline
  To describe dysphonia: from 0 (normal) to 3 (severe)
French scale "Batterie d'Evaluation Clinique de la Dysarthrie" (Clinical Evaluation of Dysarthria) phonetics characteristics | 5 minutes at baseline
  Phonetic characteristics of voice: nine items, each quoted from A (normal) to E (strongly abnormal).
French scale "Batterie d'Evaluation Clinique de la Dysarthrie" (Clinical Evaluation of Dysarthria) perceptive analysis. | 5 minutes at baseline
  To describe the clinical characteristics of dysarthria in idiopathic oromandibular dystonia. Perceptive score (min=best=0; max=worst=20)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Kreisler, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU, Lille, France